CLINICAL TRIAL: NCT03145753
Title: Impact on New HIV/HCV Infection Diagnoses and Costs of Two HIV/HCV Testing Programs "Education and Support Only" Versus "Education and Support Plus a Resourced External Program (DRIVE 03)"
Brief Title: Education vs Education Plus Intervention in HIV/HCV Diagnosis (DRIVE 03)
Acronym: DRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: PI16/00551
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2017-05

CONDITIONS: HIV Infection; HCV Coinfection
Keywords: HIV testing program; HCV testing program; education
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: DRIVE study (Diagnóstico Rápido de la Infección por VIH/HCV en España, in English Rapid HIV/HCV testing in Spain) was designed to investigate the different aspects of HIV testing. DRIVE 01 and 02 had been already completed and communicated.
  This new study has been designed as a prospective randomized clustered crossover study in one Health Care Area of Madrid Spain, to compare two implementation HIV/HCV testing programs: only EDSUP vs. EDSUP plus a resourced HIV/HCV testing program which provide rapid HIV/HCV tests, and testing staff to conduct all procedures.
  Four PCC´c belonging to the influenced area of Ramón y Cajal Area will be randomized 1:1 to receive sequentially any of the two HIV/HCV testing programs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV/HCV Education plus Testing (Experimental): In this arm education should be provided and also resources for testing, HIV/HCV rapid tests and Testing staff different from clinical practice resources
  Interventions: Other: HIV/HCV Education plus Testing
- HIV/HCV Education (Active Comparator): In this arm only education should be provided
  Interventions: Other: HIV/HCV Education

INTERVENTIONS:
Other: HIV/HCV Education plus Testing — Education included a half day educational program and the provision of supporting materials to enhance HIV testing, such as a clinical decision algorithm to perform HIV test and clinical remainders to help meet with the current Spanish Early Diagnosis HIV Testing Recommendations. Half day educational program, to promote early diagnosis of HIV, HCV, in a Primary Care Health Area.To Improve knowledge and current trends in the prevention, diagnosis and management of HIV infection among non health professionals specialists in infectious diseases.DRIVE 03 program will offer rapid HIV tests, and testing staff to conduct all study procedures.The study activities will be carried out by the trained testing staff.
  Arms: HIV/HCV Education plus Testing
Other: HIV/HCV Education — Only education and support will be provided in this arm
  Arms: HIV/HCV Education

SUMMARY:
Objectives: A targeted HIV testing strategy (TTS) through an HIV risk of exposure and indicator conditions (RE&IC) questionnaire resulted in same rate of new HIV infection diagnosis (NHID), coverage and even reduced costs compared with a universal non targeted (Non TSS) HIV testing strategy in a prior study (DRIVE 01). To compare number of New HIV/HCV Infection Diagnoses (NHID HIV/HCV) and costs two HIV/HCV testing programs in the Primary Health Care: an educational and support only initiative to enhance HIV /HCV testing (EDSUP) or EDSUP plus a resourced external program (DRIVE 03).

Methodology: Prospective, randomized 1:1, clustered, crossover study, in one Health Care Area of Madrid, Spain, comparing the implementation of two HIV testing programs, EDSUP only vs. EDSUP plus DRIVE 03 program in 4 Primary Care Centers (PCC´s). People randomized to EDSUP plus DRIVE 03 program, non HIV infected, between 18-65 years, attending to any of the 4 PCC´s, not previously included in the study will be offered to participate. HIV testing program will be evaluated by measuring absolute number of new diagnosed infections (NDI) HIV/HCV and costs. Other outcomes considered will be people assigned and offered to participate, number of HIV tests performed, coverage (HIV /HCV tests/assigned population ratio), and rate of NDI HIV/HCV per ‰ tests performed. Six months prior to randomization main outcome variables will be recorded in the 4 PPC´s. Before randomization, EDSUP will be equally implemented in the 4 PCC´s. After randomization, first six months, DRIVE 03 program will be implemented in 2 PCC´s and in the other 2 observation of interest variables will be conducted. After first 6 month study period, PCC´s will be crossover to the opposite arm of randomization. DRIVE 03 program will offer rapid HIV tests, and testing staff to conduct all study procedures. For NDI HIV/HCV, molecular epidemiology, delayed diagnosis, retention in care, HIV/HCV treatment and control/eradication will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Have attended to one of the PCC´s randomized to DRIVE 03 HIV testing program,
* Be 18-70 years
* Have understood, accept and sign the written informed consent, and in case of inability, it will be signed by the legal representative.

Exclusion Criteria:

* A prior HIV diagnosis,
* have already been included in the DRIVE 03 study,
* inability to understand the Spanish language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7989 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Number of New HIV HIV/HCV Diagnosis | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jesus Pérez Elías, MD, PhD, Principal Investigator — Hospita Camon y Cajal, IRYCIS
Locations (2):
- Spain (2):
  - Centro de Salud Garcia Noblejas, Madrid
  - Hospita Ramon y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No